

# Consent of an Adult to Be in a Research Study

In this form "you" means a person 18 years of age or older who is being asked to volunteer to participate in this study.

| Participant's Name Medical Record Number: | |
|---|---|
| Principal Investigator: | Sue Brown, MD |
| | UVA Center for Diabetes Technology |
| | Box 400888 |
| | Charlottesville, VA 22908 Telephone: (434) 982-0602 |
| Sponsor: | UVA Strategic Investment Fund |

# What is the purpose of this form?

This form will provide you with information about this research study. You do not have to be in the study if you do not want to. You should have all your questions answered before you agree to be in this study.

Please read this form carefully. If you want to be in the study, you will need to sign this form. You will be given a signed copy of this form.

# Who is funding this study?

This study is paid for by a funding from the University of Virginia Strategic Investment Fund.

# Why is this research being done?

The purpose of this study is to understand how glucose changes after having an islet transplantation (infusion of isolated islets from a donor pancreas into another person). This study is intended to help researchers understand how glucose levels change after surgery and how this information can be used in the development of automated insulin delivery systems (i.e. Artificial Pancreas Systems).

You are being asked to be in this study, because you have had an islet transplantation.

Up to 40 people will be in this study at UVA.

# How long will this study take?

Your participation in this study will require two (2) study visits over approximately 4 months. Visit 1 is a screening visit to determine your eligibility. This visit may take about 2 hours to complete. Visit 2 is a 1 hour visit to train you on the study requirements. Visit 1 and 2 may occur on the same day if you meet study eligibility. Visit 3 is for you to return the CGM equipment to the study team. This visit may occur at UVA or remotely.

 Version: 04/06/18



IRB-HSR Approval Date:27NOV2018

IRB-HSR Expiration Date: 26NOV2019



Note: All procedures, assessments and tests described in this consent are being done solely for research purposes.

# What will happen if you are in the study?

### SCREENING (visit will last about 2 hours)

Visit 1 (Day 1):

If you agree to participate, you will sign this consent form before any study related procedures take place. Before you can start in the study, there will be a screening period. You will have tests and procedures during this time to make sure you are eligible and it is safe for you to participate. These include the following:

- Collection of information about you: your diabetes history, past and current medical conditions, surgical procedures, menstrual history (females), allergies, medications and supplements, social history (including drinking, smoking and drug habits), and whether or not you have various symptoms.
- Your pump settings and/or average daily insulin use over the past seven days.
- Collection of your contact information
- Physical exam
- HbA1c test (results collected within the last four weeks is acceptable)
- Additional blood tests if your study doctor has any concerns about medical conditions that might affect your participation in the study (results collected within the last six months is acceptable)
- A urine or blood pregnancy test if you are a woman who can become pregnant. The pregnancy test
  must be negative in order for you to participate and will be repeated at each follow-up clinic visit
  during the study.

If these tests show you are eligible, you will return to the research site either that day or another day for Visit 2 to begin study treatment.

### STUDY PROCEDURES

# <u>VISIT 2 – Study Equipment Training (will take approximately 1-3 hours to complete depending on your knowledge of the continuous glucose monitor):</u>

You will receive training on the continuous glucose monitor during this visit. This will include inserting the sensor, calibrating the equipment, and caring for the insertion site. You will be instructed on how to properly obtain a blood glucose value.

Using acetaminophen-containing medications (i.e. Tylenol) may affect the performance of the continuous glucose monitor. Limited use of acetaminophen will be permitted, but you will be asked to write down when you have taken this medication. You should not use the CGM values for treatment decision for 24 hours after using acetaminophen.


# IRB-HSR#20294: Continuous Glucose Monitoring and Closed Loop Control in Islet Transplant Recipients



You will be taught how to calibrate the CGM per manufacturer's guidelines. You will be asked to perform all required calibrations with fingerstick glucose measurements. Any additional BG tests normally done by you should continue without interruption.

You will be asked to bring your personal laptop so study staff can download the app that will assist in providing the study team the CGM data (i.e. Dexcom CLARITY or diasend®). Study staff will help you set up an account and instruct you on how to download the study CGM from home.

If you use insulin injections rather than an insulin pump, you will be asked to record your insulin injections in a commercially available app such as MySugr.

You can call or visit the study team and study physician as needed. You will be given the telephone numbers of the study team so you call someone 24-hours a day.

### Data Collection Period Prior to Experimental Admission (approximately 28-90 days)

During this collection phase, the study team will collect information on your glucose values and insulin treatment. Data collection may continue up to 3 months.

During this collection phase, you will follow your usual regimen. However, we will ask that you wear the continuous glucose monitor along with your normal insulin treatment (i.e. insulin pump or multiple daily injections). You will be asked to use the bolus calculator function on your insulin pump and enter the carbohydrate information that you eat during the week. You will be asked to record any bolus insulin treatments that you have provided yourself with use of an insulin pen or needle injection.

You will be asked to download equipment and provide the data to the study team after approximately every 7 days. Study team will review this data to check that the data is being collected correctly. You may be asked to do more frequent downloads or to repeat this collection phase.

### Study Procedures that will occur during Visit 3:

You will be asked to return the study equipment. This may involve a trip to UVA or could be done remotely by mailing the devices to us with contact from the study staff. An optional HbA1c test may also be done for research purposes (less than ½ teaspoon).




### **STUDY SCHEDULE**

| Study Procedures | Screening | Study<br>Training | Data<br>Collection | Final Visit |
|---|---|---|---|---|
| Visit | 1 | | 2 | 3 |
| Days | 1 | 2 | 2-90 | 33 or 92 |
| Duration (approximate times) | 2 hours | ~1-3 hour | 28 -90 days | 1 hour |
| Location | UVA | UVA | Home | UVA or<br>Home |
| Informed Consent | Х | | | |
| Clinical exam & medical history | Х | | | |
| Inclusion/Exclusion Criteria | Х | | | |
| Screening Labs | Х | | | |
| Urine pregnancy test (women able to become pregnant) | Х | Х | | |
| CGM Use | | Х | Х | |
| Exercise | | | | |
| Equipment Downloads | | | ~Once a<br>week | Х* |

<sup>\*</sup>Post admission

### What are your responsibilities in the study?

You have certain responsibilities to help ensure your safety. These responsibilities are listed below:

- You must attend each study visit as advised by the study staff.
- You must be completely truthful about your health history.
- Follow all instructions given.
- You should tell the study doctor or study staff about any changes in your health or the way you feel.
- Answer all of the study-related questions completely.
- Inform the study doctor or study staff as soon as possible if you have to take any new medications, including anything prescribed by a doctor or those that you can buy without a prescription (over-the-counter), including herbal supplements and vitamins. The study doctor will let you know if you can take these medications.

### **Blood Testing**

We will take (or "draw") up to 6 ½ teaspoons of blood during the study.

The screening visit (6 teaspoons of blood): The blood we taken at the screening appointment will be tested to measure your diabetes control, your thyroid function, how well your kidneys/liver work, the amount of certain salts and sugars, and to see if you are pregnant (females).

Visit 3 (½ teaspoon of blood) The Hemoglobin A1c blood test.




You will take fingersticks during the trial to measure your blood glucose levels. The physician may ask that you take more fingersticks to help monitor your glucose levels. Please note that if you access LabCorp, more blood will be taken than the UVa laboratory. No other blood sampling will be completed during the trial.

When these tests are done, any left-over sample will be thrown away or they will be de-identified. This means there is no information that could be used by anyone to determine who the sample came from.

## If you want to know about the results before the study is done:

During the study, your study leader will let you know of any test results that may be important to your health. In addition, as the research moves forward, your study leader will keep you informed of any new findings that may be important for your health or may help you decide if you want to continue in the study. The final results of the research will not be known until all the information from everyone is combined and reviewed. At that time, you can ask for more information about the study results.

# What are the risks of being in this study?

Risks and side effects related to the devices include:

### Risks related to treating type 1 diabetes (with or without using study equipment)

### Likely:

- Risk of possible mild to moderate low blood sugar and possible symptoms of low blood sugar, such as sweating, trembling, difficulty thinking, dizziness, and feeling uncoordinated.
- Risk of possible mild to moderate high blood sugars and possible symptoms of high blood sugars such as thirst and frequent urination. You may have a higher level of sugar in your urine.

### Rare but serious

- Risk of severe temporary low blood sugar (hypoglycemia) that can lead to unconsciousness, hypoglycemic seizure, hospitalization or even death.
- Risk of prolonged high blood sugar leading to diabetic ketoacidosis, hospitalization, and coma. DKA can lead to renal failure (kidney failure), cardiac arrhythmia (irregular heartbeat), myocardial infarction (heart attack), rhabdomyolysis (muscle breakdown), and even death.

### Fingerstick Risks

### Likely:

- Pain at site of lancet (finger-pricking needle) use
- Bleeding at site of lancet use


# IRB-HSR#20294: Continuous Glucose Monitoring and Closed Loop Control in Islet Transplant Recipients



### Less Likely:

Incorrect information from a false low or false high fingerstick value

### Rarely:

Infection at site of lancet use

### Continuous Glucose Monitoring Sensor Risk

### <u>Likely:</u>

- Failure or lack of sensitivity of the continuous glucose monitor sensor that requires replacement / insertion of new sensor
- Fingerstick for calibration of the continuous glucose monitor
- Discomfort from insertion of sensor

### **Less Likely:**

- Bruising less than ½ inch
- Bleeding less than ¼ teaspoon
- Sensitivity to adhesives with use of continuous glucose monitor resulting in skin irritation, redness, blistering, scarring, systemic allergic reaction or secondary skin infection

### Rarely:

- Swelling or redness at insertion site
- Psychological reaction to viewing the continuous glucose monitor information or attending to continuous glucose monitor alarms or fingerstick blood glucose values.
- Breakage of the continuous glucose monitor sensor under the skin with possible symptoms of skin
  irritation and inflammation. If a sensor breaks and no portion of it is visible above the skin, do not
  attempt to remove it. Please call the study team or seek immediate medical assistance. Seek
  professional medical help if you have symptoms of infection or inflammation redness, swelling or
  pain at the insertion site.

# <u>Performing a serum (blood) or urine pregnancy tests females who are able to become pregnant):</u> <u>Less Likely:</u>

False positive or false negative results

### Risk of Sharing the Continuous Glucose Monitor

We may use the continuous glucose monitor equipment with other study subjects. The sensors will not be shared. The transmitter wirelessly sends your glucose information from the sensor to the receiver. The transmitter, which snaps into the sensor, will be cleaned thoroughly with a diluted mixture of bleach or another appropriate cleaner after use. The FDA approved the continuous glucose monitor as a 'single use device'. This means that they recommend that only one person use this device as there is a rare risk that a blood borne pathogen, such as Hepatitis B, may be spread if used with multiple patients.




### **Blood Donation**

If you participate in this study, it may affect your ability to donate blood. If you have any questions, call the organization where you donate blood and talk to one of their nurses.

### Risks of having your blood drawn:

Having blood drawn may cause:

- ✓ pain (common),
- ✓ a bruise (sometimes),
- √ fainting or passing out (not very often), and
- ✓ infection (rare).

If the people doing the study are exposed to your blood or body fluids in a way that could give them a disease, your blood may be tested. The tests might check for:

- ✓ hepatitis,
- ✓ HIV (Human Immunodeficiency Virus), or
- ✓ other infections.

You and the person exposed would be told the test results. However, your name would be kept private. If your test is positive for hepatitis or HIV or any other infection that may affect your clinical care, we will tell you the results and help you understand what the results mean for you.

### Risks for women:

Being in this study might hurt your unborn baby, so you will not be able to join or stay in the study if you are pregnant. You must use an effective method of birth control during the study. If you are pregnant now, or get pregnant during the study, please tell us right away.

### Other unexpected risks:

You may have side effects that we do not expect or know to watch for now. Call the study leader if you have any symptoms or problems.

# Could you be helped by being in this study?

You will not benefit from being in this study. However, the information researchers get from this study may help others in the future.

# What are your other choices if you do not join this study?

You do not have to be in this study to be treated for your illness or condition. You can get the usual treatment for your T1DM even if you choose not to be in this study. The usual treatment would include continuing your home insulin regimen.


### IRB-HSR#20294: Continuous Glucose Monitoring and Closed Loop Control in Islet Transplant Recipients



However, in order to do this study we must change the equipment that you use in usual treatment. This would be wearing the study CGM.

- o If you are a patient at UVa, your usual care will not be affected if you decide not to participate in this study.
- o If you are an employee of UVa your job will not be affected if you decide not to participate in this studv.
- o If you are a student at UVa, your grades will not be affected if you decide not to participate in this study.

# Will you be paid for being in this study?

You will be paid for participating in the study. You will receive payment after the study equipment has been returned to the study team. You should get your payment by check about 4 weeks after finishing the study. The income may be reported to the IRS as income.

- Completion of Visit 2 (Study equipment training): \$100
- o Completion of Visit 3 (Data Collection Period): \$50/month up to 3 months (total \$150)

If you do not finish the study, you will be paid for the visits that you completed. If the study leader says you cannot continue, you will be paid the full amount for the study.

You will receive reimbursement for travel in the following way:

- If greater than 50 miles from the Center, mileage will be paid at the current state rate per mile, up to a maximum of 500 miles
- If greater than 200 miles from the Center, you may be compensated for air travel up to the rate of \$500 round trip
- Hotel compensation up to \$150/night with a maximum stay of one night if traveling more than 150 miles from the Center
- Study subject traveling by air travel will be compensated for up to 2 days of meals at \$69/day.
- Study subjects traveling by air travel, a taxi trip to and from the Charlottesville airport and UVA will be compensated at \$25/trip with a maximum of 2 trips.
- Study subjects traveling by air travel will be compensated for up to 2 days of airport parking of \$10/day with a maximum of 2 days.

If you pay for your own travel, receipts will be required to obtain reimbursement.

If you owe money to any Virginia state agency, the state can use the money you earn in this study to pay those debts. These state agencies include the UVa Medical Center, VCU Medical Center or a college or university. The money may be withheld to pay back debt for such things as unpaid medical bills, taxes, fines, child support. Even if this happens, the money you earn may be reported to the IRS as taxable income.




# Will being in this study cost you any money?

All of the procedures in this study will be provided at no cost to you or your health insurance. You will be responsible for using your own insulin pump, insulin and glucometer. Parking is available at no cost at the research site.

You and/or your insurance company must pay for any tests or care given beyond what is required in this study. In addition, you and/or your health insurance may also have to pay for other drugs or treatments that are given to help you control any side effects. You will have to pay for any costs not covered by your health plan. You may be responsible for any co-payments or deductibles. You may wish to ask your insurance company for an estimate of what these costs might be or if pre-approval is required.

# What if you are hurt in this study?

You do not give up any legal rights, such as seeking compensation for injury, by signing this form. If you feel you have been injured as a result of this study you may contact the Principal Investigator or the IRB (phone numbers are located near the end of this form). If you are hurt as a result of being in this study, there are no plans to pay you for medical expenses, lost wages, disability, or discomfort. The charges for any medical treatment you receive will be billed to your insurance. You will be responsible for any amount your insurance does not cover.

# What happens if you leave the study early?

You can change your mind about being in the study any time. You can agree to be in the study now and change your mind later. If you decide to stop, please tell us right away. You do not have to be in this study to get services you can normally get at the University of Virginia.

Even if you do not change your mind, the study leader can take you out of the study. Some of the reasons for doing so may include

- a) Your study physician is concerned about your health
- b) Your condition gets worse
- c) The side effects of the treatment are too dangerous for you
- d) New information shows the treatment will not work or is not safe for you
- e) You do not follow your doctor's instructions
- f) The study sponsor closes the study for safety, administrative or other reasons
- g) If you become pregnant during the study
- h) If the study physician is concerned about the frequency of acetaminophen use during the study

If you decide to stop being in the study, we ask that you notify the research team so any scheduled admissions may be cancelled. The CGM and activity tracker study equipment remain property of the CDT and will need to be returned.



# How will your personal information be shared?

The UVa researchers are asking for your permission to gather, use and share information about you for this study. If you decide not to give your permission, you cannot be in this study, but you can continue to receive regular medical care at UVA.

# If you sign this form, we may collect any or all of the following information about you:

- o Personal information such as name, address and date of birth
- Social Security number ONLY IF you are being paid to be in this study
- Your health information if required for this study. This may include a review of your medical records and test results from before, during and after the study from any of your doctors or health care providers. This may include mental health care records, substance abuse records, and/or HIV/AIDS records.

### Who will see your private information?

- The researchers to make sure they can conduct the study the right way, observe the effects of the study and understand its results
- People or groups that oversee the study to make sure it is done correctly
- o The sponsor(s) of this study, and the people or groups it hires to help perform or review this research
- Insurance companies or other organizations that may need the information in order to pay your medical bills or other costs of your participation in the study
- Tax reporting offices (if you are paid for being in the study)
- People who evaluate study results, which can include sponsors and other companies that make the drug or device being studied, researchers at other sites conducting the same study, and government agencies that provide oversight such as the Food and Drug Administration (FDA) if the study is regulated by the FDA.
- o If you tell us that someone is hurting you, or that you might hurt yourself or someone else, the law may require us to let people in authority know so they can protect you and others.

Some of the people outside of UVa who will see your information may not have to follow the same privacy laws that we follow. They may release your information to others, and it may no longer be protected by those laws.

The information collected from you might be published in a medical journal. This would be done in a way that protects your privacy. No one will be able to find out from the article that you were in the study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.




# What if you sign the form but then decide you don't want your private information shared?

You can change your mind at any time. Your permission does not end unless you cancel it. To cancel it, please send a letter to the researchers listed on this form or complete the "Leaving the Study Early" part of this form and return it to the researchers. Then you will no longer be in the study. The researchers will still use information about you that was collected before you ended your participation.

A copy of this consent form will be put in your medical record. (This is not the same as the record of this research study.) This means that everyone who is allowed to see your medical records will be able to find out that you are in this study. This is done so your regular doctors will know what you receive as part of this study. If you have other health problems during the study, they will be able to treat you properly.

### Please contact the researchers listed below to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

### **Principal Investigator:**

Sue Brown, MD UVA Center for Diabetes Technology Box 400888 Charlottesville, VA 22903 Telephone: (434) 982-0602

# What if you have a concern about this study?

You may also report a concern about this study or ask questions about your rights as a research subject by contacting the Institutional Review Board listed below.

University of Virginia Institutional Review Board for Health Sciences Research PO Box 800483 Charlottesville, Virginia 22908

Telephone: 434-924-9634

When you call or write about a concern, please give as much information as you can. Include the name of the study leader, the IRB-HSR Number (at the top of this form), and details about the problem. This will help officials look into your concern. When reporting a concern, you do not have to give your name.


| IRB-HSR#20294: Continuous Glucose Monitoring and Closed Loop Control in Islet Transplant Recipients | | |
|---|---|---|
| Signatures | | |
| What does your signature mea | | |
| | | is study that is not clear to you. Your |
| | | all your questions have been answered. If |
| you sign the form, it means that | t you agree to join the study. You w | ill receive a copy of this signed document. |
| Consent From Adult | | |
| PARTICIPANT | PARTICIPANT | DATE |
| (SIGNATURE) | (PRINT) | DATE. |
| To be completed by participant | | |
| Person Obtaining Consent | | |
| By signing below, you confirm tl | nat you have fully explained this stud | dy to the potential subject, allowed them |
| time to read the consent or hav | e the consent read to them, and hav | ve answered all their questions. |
| PERSON OBTAINING CONSENT | PERSON OBTAINING CONSENT | DATE |
| (SIGNATURE) | (PRINT) | -··· <u>-</u> |
| Notification of My Heal | th Caro Providor | |
| | · | |
| rour nealth care provider will be | e notified of your participation in this | s study. |
| Please indicate helow whether y | you want us to notify your hoalth car | re provider that you have agreed to take |
| part in this study. | want us to notify your nearth car | e provider that you have agreed to take |
| , | to a second second | |
| study. | doctor to notify my health care prov | ider that I have agreed to take part in this |
| • | | |
| Health Care Provider Name: | | |

\_\_\_\_\_ No, I do not want the study doctor to notify my health care provider that I have agreed to take part


**Health Care Provider Address:** 

in this study or I do not have a health care provider.

Study team will send a copy of the consent form to the health care provider.

# IRB-HSR#20294: Continuous Glucose Monitoring and Closed Loop Control in Islet Transplant Recipients Leaving the Study Early Signatures should be obtained in this section if you decide to leave the study early.

If you leave the study early the study leader will keep the data collected about you up until the time you leave the study to help determine the results of the study. Check one option below:  $_{\perp}$  I am withdrawing my consent from the intervention or treatment part of this study but agree to continue to have follow up information about me collected by the study team. The follow up information will be collected by: <INSERT APPLICABLE OPTIONS> Phone call within 36 hours after the hotel admission discharge. I am withdrawing my consent for this study. No additional information may be collected about me including follow up information from my medical records. **Consent from Adult** PARTICIPANT **PARTICIPANT** DATE (SIGNATURE) (PRINT) To be completed by participant if 18 years of age or older. **Person Obtaining Consent** By signing below you confirm that you have fully explained this study to the potential subject, allowed them time to read the consent or have the consent read to them, and have answered all their questions. PERSON OBTAINING CONSENT PERSON OBTAINING DATE

CONSENT (PRINT)

(SIGNATURE)